CLINICAL TRIAL: NCT01425086
Title: Clinical Performance of the Embrace Isothermal Mattress in Stabilizing Temperatures of the Preterm Infants During Thermal Weaning
Brief Title: Clinical Performance of the Embrace Isothermal Mattress
Acronym: KBW
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Vinod K. Bhutani, Professor of Pediatrics, Stanford University
Other Study IDs: SU-03222011-7607; eProtocol 19750 (Other: Stanford University)
Record Dates: First submitted 2011-08-24; First posted 2011-08-29 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Hypothermia
Keywords: Incubator,; hypothermia,; preterm,; low-birthweight infants,; embrace device,; phase change materials; PCM
MeSH Terms: conditions — Hypothermia; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Incubator temperature support: Infant will be cared for in the current ongoing policy-driven temperature support provided by the incubator and handling as per bedside nursing interventions. Infant will be followed clinically until discharge from Lucile Packard Hospital (average 4 weeks).
  Interventions: Device: Embrace, PCM, warming blanket
- Embrace blanket warming: Infant will be placed and wrapped in the embrace blanket and cared for and monitored for temperature support and monitored by bedside nursing interventions, as needed. Infant will be followed clinically until discharge from Lucile Packard Hospital (average 4 week
  Interventions: Device: Embrace, PCM, warming blanket

INTERVENTIONS:
Device: Embrace, PCM, warming blanket — Infant will be placed on a blanket that encloses the Embrace device, The infant will be wrapped in this blanket to create a snug, comfortable and warm "micro-environment".
  Other Names: Embrace Device; Embrace Isothermal Mattress; Embrace Blanket; PCM blanket

SUMMARY:
The purpose of this pilot study is to evaluate the performance of a new warming technology (Embrace Isothermal Mattress) during the thermal weaning of premature infants from incubators to open cribs. The investigators aim to study the Embrace Isothermal Mattress over a 24-hour period before the infant is transitioned out of the incubator.

DETAILED DESCRIPTION:
The investigators aim to use the results of this pilot study in preparation for a larger, longer, multi-center clinical trial testing the performance of the Embrace Isothermal Mattress during the weaning of premature infants from incubators to open cribs (thermal weaning). Specifically, this study would provide physiological data (e.g. temperature, weight) and operational experience (e.g. logistical issues, familiarity with technology) that would assess the short-term effectiveness (< 24 hours) of the new technology in maintaining temperature stability as well as informing the subsequent trial.

This study will build upon two primary bodies of scientific knowledge: (1) the applicability of an isothermal mattress as a supplemental heat source during thermal weaning and (2) basic clinical knowledge of the quality, quantity, and timing of warming during the thermal weaning process.

First, current thermal weaning processes at LPCH are heavily dependent upon prolonged use of incubators. Additional sources of warming include radiant warmers, transwarmers (e.g. one-time use gel-packs), skin-to-skin contact (e.g. Kangaroo Mother Care), and others. While all provide sufficient warming during thermal weaning but are not always ideal (e.g. incubators separate mother and baby, radiant warmer and transwarmers have varying abilities to stabilize temperature over prolonged periods, and skin-to-skin contact is not constantly available). In contrast, the Embrace Isothermal Mattress is based on a wax-like phase-change-material (PCM) that allows for an extremely stable long-term heat exchange with an infant. It was designed to function without a constant source of electricity and is relatively portable allowing for its use as a supplement to incubators, skin-to-skin contact, and other warming techniques.

Secondly, this study will inform future clinical practices specifically in thermal weaning and generally in neonatal temperature regulation. Thermal weaning occurs when the incubator's set temperature is incrementally lowered by nurses in preparation for a transition to an open crib. Eventually, a clinical decision is made to clothe the infant and turn off the incubator (based upon physiological markers and nursing experience). A period of observation of the clothed infant within the switched-off incubator (immediate to 12 hours based on a survey of LPCH nurses) then precedes transition to an open crib. A series of retrospective chart reviews has observed a range of thermal weaning practices between and within LPCH-affiliated nurseries possibly due to a wide interpretation of existing thermal weaning protocols (e.g. weaning at different post- menstrual ages, physiological characteristics, cognitive development). The investigators are hopeful that this study will provide additional scientific data to inform clinical decision-making during thermal weaning.

Ultimately, the research performed in this pilot study and subsequent clinical trial will determine whether the Embrace Isothermal Mattress may facilitate a more optimal transition of an infant from an incubator to an open crib. For example, if infants are found to transition effectively at lower body weight and post-menstrual age while still maintaining temperature stability while using the Embrace Isothermal Mattress, then clinicians can offer an alternative thermal weaning method with additional secondary benefits. Specifically, this early transition may facilitate earlier mother-child bonding and improve the infant's quality of life ultimately leading to a more advanced developmental stage upon discharge from the PICN. In addition, use of this new technology as an alternative for weaning may free incubators for more life-threatening cases, ultimately providing for more efficient and cost-effective use of PICN resources. Therefore, the end goal is to improve overall clinical practice and patient experience by introducing and evaluating a potentially beneficial warming technology.

ELIGIBILITY:
Inclusion Criteria:

1. Prematurity (27 to 34 weeks post-menstrual age at birth, 33 to 35 weeks post-menstrual age at screening)
2. At risk for environmental hypothermia
3. Cared for in an incubator
4. Currently undergoing thermal weaning (no less than 72 hours prior to anticipated thermal weaning to transition to an open crib)
5. Cardio-respiratory stability (as determined by physician/NNP)
6. Written informed parental consent

Exclusion Criteria:

1. Continuing requirement of phototherapy
2. Continuing requirement of assisted ventilation (e.g. CPAP)
3. Cardio-respiratory instability (as determined by physician)
4. Clinically-significant congenital abnormalities (as determined by PI)
5. Acidosis or ongoing sepsis
6. Dehydration (defined by hypernatremia with serum sodium > 150 meq/L)
7. Any additional concurrent high risk medical/surgical condition (as determined by physician, NNP or PI)
8. Refusal of participation by parents -

Ages: 1 Day to 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Low birth weight neonates
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12-20 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Temperature Stability | 48 hours
  As monitored by ambient (environmental) temperature, infant's core and surface temperature

SECONDARY OUTCOMES:
Safety assessment by absence of change in cardio-respiratory events | 48 hours
  As monitored by heart rate, respiratory rates, pulse-oximetry and occurrence of apnea events

CONTACTS AND LOCATIONS:
Overall Officials: Vinod K. Bhutani, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States